CLINICAL TRIAL: NCT07194668
Title: Immunogenicity of a Fractional Adult Dose of the Malaria Vaccine R21/Matrix-M - A Noninferiority Trial
Brief Title: R21/MM Dosing, Presentations, and Preservatives
Acronym: VAC100
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: University of Oxford (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: MAL25005
Record Dates: First submitted 2025-09-02; First posted 2025-09-26 (Actual); Last update posted 2026-01-12 (Actual); Status verified 2025-08

CONDITIONS: Plasmodium Falciparum Malaria; Malaria; Vaccine Reaction
Keywords: Plasmodium Falciparum Malaria; Malaria Vaccine
MeSH Terms: conditions — Malaria, Falciparum; Malaria

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- The standard adult vaccine dose (Active Comparator): Adults and adolescents receiving the standard adult vaccine dose
  Interventions: Biological: 10μg R21/50μg Matrix-M
- A half of the standard adult vaccine dose with adaptor Preservative Free (Active Comparator): Adults and adolescents receiving a half of the standard adult vaccine dose with adaptor Preservative Free (n=125)
  Interventions: Biological: 5μg R21/50μg Matrix-M with adaptor preservative free
- A half of the standard adult vaccine dose with 2PE Preservative (Active Comparator): Adults and adolescents receiving a half of the standard adult vaccine dose with 2PE Preservative (n=125)
  Interventions: Biological: 5μg R21/50μg Matrix-M with 2PE preservative

INTERVENTIONS:
Biological: 10μg R21/50μg Matrix-M — Adults and adolescents receiving the standard adult vaccine dose: 10μg R21/50μg Matrix-M (n=125)
  Arms: The standard adult vaccine dose
Biological: 5μg R21/50μg Matrix-M with adaptor preservative free — Adults and adolescents receiving a half of the standard adult vaccine dose: 5μg R21/50μg Matrix-M using two presentations: 10 dose vials with adaptor Preservative Free (n=125)
  Arms: A half of the standard adult vaccine dose with adaptor Preservative Free
Biological: 5μg R21/50μg Matrix-M with 2PE preservative — Adults and adolescents receiving a half of the standard adult vaccine dose: 5μg R21/50μg Matrix-M using two presentations: 10 dose vials with 2PE Preservative (n=125)
  Arms: A half of the standard adult vaccine dose with 2PE Preservative

SUMMARY:
This is a single blind randomised controlled trial. This study aims to assess whether a half-dose of the R21/Matrix-M malaria vaccine is as effective as the full dose in child and adults. The results will help optimize vaccine usage and improve malaria prevention strategies.

All participants will receive the same number of injections and will be randomly assigned to receive one of the followings:

1. The standard dose (10μg R21/50μg Matrix-M) of the malaria vaccine is administered in three doses over a two-month period (at Month 0, 1, and 2), followed by a booster dose at Month 11 (n=125).

   or
2. A half dose (5μg R21/50μg Matrix-M) of the malaria vaccine is administered in three doses over a two-month period (at Month 0, 1, and 2), followed by a booster dose at Month 11.

If participant receive the half dose, it will come from one of two types of vaccine:

2a. 10 dose vials with adaptor Preservative Free (n=125) 2b. 10 dose vials with 2PE Preservative (n=125)

Clinical procedure for participants:

* Standardized symptom questionnaire
* Physical examination:

  * Weight, height, pulse, blood pressure, respiratory rate, tympanic temperature.
  * Spleen and liver size will be recorded if palpable.
  * Pregnancy test (for female of child bearing potential)
* Venous blood collection (Pre-vaccination) 3mL
* Vaccination

ELIGIBILITY:
Inclusion Criteria:

* Residence in a study village for the study period, i.e. 12 months.
* Age 14 years to 60 years.
* Written informed consent/assent provided by participants (or a parent/guardian in case the participant is under 18 years old).

Exclusion Criteria:

* Pregnancy, plan to get pregnant within one month of vaccination, or breastfeeding.
* Acute illness requiring intervention.
* A history of an adverse reaction to study vaccine.
* Prior receipt of any other malaria vaccine.
* Enrolment in another intervention trial in the last month.
* Planned enrolment in another intervention trial in the coming 12 months.
* Regular use of Immunomodulating drugs e.g, Steroid, Methotrexate, Immunotherapy etc. in the past month and/or planned for the coming 12 months.

Ages: 14 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 375 (Estimated)
Dates: Start 2026-03-01 (Estimated); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
The concentration of antibodies against Plasmodium falciparum circumsporozoite (anti-NANP total IgG antibody) | One month after the completion of the third dose (at M3), and one month after the booster dose (at M12).
The concentration of antibodies against Plasmodium falciparum circumsporozoite (anti C-Term, and full length R21 total IgG antibody), in addition to total IgG against Hepatitis B surface antigen | One month after the completion of the third dose (at M3), and one month after the booster dose (at M12).

SECONDARY OUTCOMES:
Adverse event and severe adverse event reports for safety and tolerability assessment of the standard adult vaccine dose 10μg R21/50μg Matrix-M and a half of the standard adult dose 5μg R21/50μg Matrix-M | At Month 1, Month 2, Month 3, Month 11 and Month 12
Adverse event and severe adverse event reports for safety and tolerability assessment a half of the standard adult dose 5μg R21/50μg Matrix-M with 2PE preservative vs, without 2PE preservative. | At Month 1, Month 2, Month 3, Month 11 and Month 12

OTHER OUTCOMES:
Assays to assess presence or absence of other factors potentially affecting vaccine immunogenicity | Month 0, Month 3, Month 11 and Month 12

CONTACTS AND LOCATIONS:
Locations (2):
- Bangladesh (2):
  - Lama Upazila Health Complex, Lāma, Lama
  - Alikadam Upazila Health Complex, Bāndarban

IPD SHARING:
Plan to Share IPD: Yes
With participant's consent, participant's data and results from blood analyses stored in the database may be shared according to the terms defined in the MORU data sharing policy (https://www.tropmedres.ac/units/moru-bangkok/bioethics-engagement/data-sharing/moru-tropical-network-policy-on-sharing-data-and-other-outputs)with data repositories such as the WorldWide Antimalarial Resistance Network (WWARN, terms of submission here: http://www.wwarn.org/tools-resources/terms-submission) or other researchers to use in the future. All personal information will be anonymised so that no individual can be identified from their treatment records, through interviews, or from mapping data.
Supporting Information: ICF, CSR